CLINICAL TRIAL: NCT04342923
Title: Early POstoperative BIomarkers in PancreatoDuodenectomy as Predictors of Complications: a Spanish Nationwide Multicentric Validation Study
Brief Title: Early POstoperative BIomarkers in PancreatoDuodenectomy: a Spanish Nationwide Study
Acronym: EPOBIPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Mario Rodriguez-Lopez, General and Digestive Surgeon, MD, PhD, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 20-1679
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Pancreaticoduodenectomy
Keywords: PANCREATICODUODENECTOMY; COMPLICATIONS; PANCREATIC FISTULA; SCORE; BIOMARKERS
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complete cohort: All patients undergoing PD during study period in all participating center/units in Spain.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Blood analysis

SUMMARY:
AIMS: To recruit a large nationwide Spanish series in order to register PF rate and other common morbidity after PD, and to perform external validation of the aforementioned score, as well as to analyze other postoperative blood parameters and biomarkers associated with complications.

METHODS: Observational prospective and multicentric cohort study to perform external validation of the above-mentioned score. All Spanish centers/units performing PD are invited to include participants. Patients will be consecutively recruited during an 8-10 months period, regardless of their annual volume of pancreatic surgery.

Study variables will be hemogram parameters on POD1 and POD2 (specifically lymphocytes), other parameters and biomarkers (RCP, lactate, procalcitonin, amylase, lipase, albumin) and the common variables concerning PD studies.

LIMITATIONS: Heterogeneity in perioperative management and in blood analysis measuring since this is a multicenter study. Possibility of underestimating the PF rate in patients without surgical drainage. Finally, the cases of mini-invasive approach or pancreatogastrostomy will receive a specific subgroup analysis since the score was designed on a series of open PD and pancreatojejunostomy.

DETAILED DESCRIPTION:
BACKGROUND: Complications after pancreatoduodenectomy (PD) are common and pancreatic fistula (PF) is among the most relevant ones. There are few studies analyzing blood parameters determined in the early postoperative period which behave as morbidity predictors. One of them defined a new and simple prognostic score based on lymphocytes count on the first postoperative day (POD1) and reactive C protein (RCP) on POD2. The internal validation statistics of the score designed in the mentioned work were satisfactory. However, that score was described in a short unicentric series

EXPECTED SAMPLE SIZE: Expected sample size is approximately 500 patients, which will show error <7.2% (with 95% confidence) for estimation score´s sensitivity and specificity. We have assumed that the PF rate is around 30%.

QUALITY CONTROL: The STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) guidelines for the correct communication and publication of observational studies will be followed. Likewise, in order to validate the aforementioned score, Transparent Reporting of a Multivariable Prediction Model for Individual Prognosis or Diagnosis (TRIPOD) will be added. The only expected failure of the 20 items that compose the TRIPOD is 6b ("notify the actions for masking the analysis"), since it is not applicable in our case.

The inclusion of patients operated on with a mini-invasive approach (laparoscopic or robotic) or the use of other anastomoses (pancreatogastrostomy) or reconstruction (Roux-en-Y) differs from the technique used in the series with which the score was originally defined (allof them, open PD with pancreato-jejunostomy and, mostly part, tutored ducto-mucosal suture and Child's single loop reconstruction). If discrepancies are detected, the corresponding subgroup analysis will be performed. Cases of conversion from a mini-invasive to open approach will be counted as such (intention-to-treat analysis).

ELIGIBILITY:
Inclusion Criteria:

* benign or malignant condition requiring surgical treatment by PD.
* Signing the informed consent form

Exclusion Criteria:

* Intra-operative findings of unresectability (pancreatic resection not be completed or palliative procedure performed)
* Other types of pancreatic resection (enucleations, distal and total pancreatectomies), as well as multivisceral resective procedures.
* Intraoperative radiotherapy
* ASA IV patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PD in Spain
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula rate | 90 days since PD
  Pancreatic fistula including biochemical, grade B and grade C according to ISGPS updated criteria 2016

SECONDARY OUTCOMES:
Clinically relevant pancreatic fistula | 90 days since PD
  Pancreatic fistula including grade B and grade C according to ISGPS updated criteria 2016
Overall complications | 90 days since PD
  Presence of any kind of complications including grades I to V according to Dindo-Clavien Classification
Severe morbidity | 90 days since PD
  Presence of any kind of complications including grades IIIa to V according to Dindo-Clavien Classification
Mortality | 90 days since PD
  Patient´s death
Comprehensive Complication Index | 90 days since PD
  Postoperative morbidity index (0-100 points) obteined by using formula described by Slankamenac et al Ann Surg 2013

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rodriguez-Lopez, MD, PhD, Principal Investigator — Hospital Clinico Universitario de Valladolid (España)
Locations (1):
- Hospital Clinico Universitario, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodriguez-Lopez M, Tejero-Pintor FJ, Bailon-Cuadrado M, Barrera-Rebollo A, Perez-Saborido B, Pacheco-Sanchez D. Impaired immune reaction and increased lactate and C-reactive protein for early prediction of severe morbidity and pancreatic fistula after pancreatoduodenectomy. Hepatobiliary Pancreat Dis Int. 2020 Feb;19(1):58-67. doi: 10.1016/j.hbpd.2019.05.003. Epub 2019 May 20. PMID 31153788